CLINICAL TRIAL: NCT01217697
Title: An Open Label Study of Abiraterone Acetate in Subjects With Metastatic Castration-Resistant Prostate Cancer Who Have Progressed After Taxane-Based Chemotherapy
Brief Title: Study of Abiraterone Acetate in Patients With Advanced Prostate Cancer
Status: Approved for marketing | Type: Expanded Access
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR017479; 212082PCR3001 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.); 2010-021425-13 (EudraCT Number)
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Prostate Neoplasms; Genital Neoplasms, Male; Urogenital Neoplasms; Genital Diseases, Male
Keywords: Metastatic Castration-Resistant Prostate Cancer (CRPC); Abiraterone Acetate
MeSH Terms: conditions — Prostatic Neoplasms; Genital Neoplasms, Male; Urogenital Neoplasms; Genital Diseases, Male | interventions — Abiraterone Acetate

INTERVENTIONS:
Drug: Abiraterone Acetate — Abiraterone acetate, type=equal, unit=mg, number=250, form=tablet, route=oral use, 4 tablets once daily.
Drug: Prednisone\Prednisolone — Participants will receive prednisone 5 mg twice daily as oral tablet OR prednisolone 5 mg (if prednisone is not available).

SUMMARY:
The purpose of this study is to collect additional safety information on abiraterone acetate administered with prednisone to patients with metastatic castration-resistant prostate cancer (CRPC).

DETAILED DESCRIPTION:
This is a study to collect information on adverse events (side effects) that occur during treatment with abiraterone acetate in patients with metastatic castration-resistant prostate cancer (CRPC). To participate in this study patients must have failed 1 or 2 chemotherapy regimens (1 of which contained a taxane such as docetaxel), reside in an area where abiraterone acetate is not yet available through local healthcare providers, and not be eligible for enrollment in any other ongoing clinical research study of abiraterone acetate. CRPC is progressive form of prostate cancer where the cancer cells become resistant to hormonal therapies that are designed to block the release or uptake of testosterone and the cancer cells metastasize (ie, spread to other parts of the body). Abiraterone acetate (referred to as abiraterone) is a drug currently under development for use in treating men with CRPC. Patients will be treated with abiraterone and prednisone daily until progression of clinical disease (ie, includes signs of clinical disease progression and/or clinical disease progression confirmed by radiographic and prostate-specific antigen [PSA] test results). Other reasons for discontinuation of treatment may include adverse events reported, initiation of other anticancer therapies, or the patient's inability to comply with dosing instructions. Patients will be followed for 30 days after the discontinuation of treatment with abiraterone acetate. Patients will take four 250-mg tablets of abiraterone orally at least 1 hour before a meal or 2 hours after a meal any time up to 10 pm every day. Patients will also take 5 mg of oral prednisone, twice daily. Each treatment cycle consists of 28 days and patients will take abiraterone continually on a daily basis until disease progression is observed at which time abiraterone will be discontinued and the dose of prednisone reduced if clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed prostate cancer
* Prostate cancer progression after previous chemotherapy as assessed by the investigator
* Received at least 1 but not more than 2 chemotherapy regimens for metastatic CRPC (at least one regimen must have contained a taxane such as docetaxel)
* Serum testosterone of less than 50ng/dL (less than 2.0 nM)
* Eastern Cooperative Oncology Group (ECOG) performance status of <=2 (ie, patients who do not have symptoms of prostate cancer and who are fully active, patients who have symptoms but are able to perform light work, or patients who are able to get around and are capable of taking care of themselves but are unable to carry out any work activities)

Exclusion Criteria:

* Serious or uncontrolled co-existent non-malignant disease (including active and uncontrolled infection)
* Active or symptomatic viral hepatitis or chronic liver disease or any abnormal liver function assessed by liver function tests
* Clinically significant heart disease as assessed by the Investigator or uncontrolled hypertension (systolic blood pressure >=160 mmHg or diastolic blood pressure >=95 mmHg)
* History of gastrointestinal disorders that may interfere with the absorption of the study drug or history of pituitary or adrenal dysfunction
* Known brain metastasis (ie, spread of cancer to the brain)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (297):
- United States (157):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Chandler, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Bellflower, California
  - Berkeley, California
  - Beverly Hills, California
  - Duarte, California
  - Encinitas, California
  - Glendale, California
  - Greenbrae, California
  - La Jolla, California
  - Laguna Hills, California
  - Long Beach, California
  - Los Angeles, California
  - Marina del Rey, California
  - Rancho Mirage, California
  - San Diego, California
  - San Francisco, California
  - Santa Rosa, California
  - Stanford, California
  - Aurora, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Fort Collins, Colorado
  - Littleton, Colorado
  - Hartford, Connecticut
  - Manchester, Connecticut
  - New Britain, Connecticut
  - Norwalk, Connecticut
  - Norwich, Connecticut
  - Southington, Connecticut
  - Stamford, Connecticut
  - Torrington, Connecticut
  - Trumball, Connecticut
  - Washington D.C., District of Columbia
  - Boca Raton, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Gainesville, Florida
  - Miami, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Palm Beach Gardens, Florida
  - Port Saint Lucie, Florida
  - South Miami, Florida
  - Atlanta, Georgia
  - Savannah, Georgia
  - Honolulu, Hawaii
  - Post Falls, Idaho
  - Chicago, Illinois
  - Decatur, Illinois
  - Harvey, Illinois
  - Niles, Illinois
  - Peoria, Illinois
  - Urbana, Illinois
  - Fort Wayne, Indiana
  - Lafayette, Indiana
  - Merrillville, Indiana
  - Muncie, Indiana
  - Bettendorf, Iowa
  - Westwood, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Marrero, Louisiana
  - New Orleans, Louisiana
  - Bangor, Maine
  - Scarborough, Maine
  - Easton, Maryland
  - Rockville, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Dearborn, Michigan
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - Lansing, Michigan
  - Rochester, Minnesota
  - Saint Louis Park, Minnesota
  - Saint Joseph, Missouri
  - Billings, Montana
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Hooksett, New Hampshire
  - Portsmouth, New Hampshire
  - Cherry Hill, New Jersey
  - Hackensack, New Jersey
  - Livingston, New Jersey
  - Morristown, New Jersey
  - New Brunswick, New Jersey
  - Paramus, New Jersey
  - Los Alamos, New Mexico
  - Albany, New York
  - Binghamton, New York
  - Brooklyn, New York
  - Buffalo, New York
  - Cooperstown, New York
  - Dunkirk, New York
  - East Setauket, New York
  - East Syracuse, New York
  - Fresh Meadows, New York
  - Glens Falls, New York
  - Mount Kisco, New York
  - New Hyde Park, New York
  - New York, New York
  - Rochester, New York
  - Stony Brook, New York
  - Syracuse, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Greenville, North Carolina
  - Hendersonville, North Carolina
  - High Point, North Carolina
  - Huntersville, North Carolina
  - Pinehurst, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Elyria, Ohio
  - Massillon, Ohio
  - Middletown, Ohio
  - Sandusky, Ohio
  - Bethany, Oklahoma
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Philadelphia, Pennsylvania
  - West Reading, Pennsylvania
  - Providence, Rhode Island
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Greenville, South Carolina
  - Myrtle Beach, South Carolina
  - Bristol, Tennessee
  - Chattanooga, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Galveston, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Temple, Texas
  - The Woodlands, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Hampton, Virginia
  - Newport News, Virginia
  - Norfolk, Virginia
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Australia (25):
  - Adelaide
  - Bedford Park
  - Box Hill
  - Camperdown
  - Footscray
  - Garran
  - Geelong
  - Heidelberg
  - Herston
  - Hobart
  - Kogarah
  - Kurralta Park
  - Liverpool
  - Nedlands
  - Port Macquarie
  - Randwick
  - South Brisbane
  - Southport Qld
  - Subiaco
  - Sydney
  - Tamworth
  - Wahroonga
  - Westmead
  - Wodonga
  - Woolloongabba
- Brazil (7):
  - Belo Horizonte
  - Curitiba
  - Porto Alegre
  - Recife
  - Rio de Janeiro
  - Salvador
  - São Paulo
- Canada (14):
  - Kelowna, British Columbia
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - Kingston, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Regina, Saskatchewan
  - Calgary
  - London
  - N/a N/a
- Colombia (6):
  - Bogotá
  - Floridablanca
  - Medellín
  - Montería
  - Pereira
  - Valledupar
- Croatia (2):
  - Split
  - Zagreb
- Czechia (5):
  - Brno
  - Hradec Králové
  - Olomouc
  - Prague
  - Ústí nad Labem
- Denmark (3):
  - Aarhus
  - Copenhagen Ø
  - Köpenhamn Ö
- Greece (6):
  - Athens
  - Athens Attica
  - Crete
  - Larissa
  - Pátrai
  - Thessalonikis
- Hong Kong (3):
  - Hong Kong
  - New Territories
  - Shatin
- Hungary (2):
  - Budapest
  - Zalaegerszeg-P Zva N/A
- Jakarta, Indonesia
- Malaysia (4):
  - Jalan Cheras N/A
  - Kota Kinabalu
  - Kuala Lumpur
  - Subang Jaya
- Mexico (13):
  - Acapulco, Guerrero
  - Aguascalientes
  - Chihuahua City
  - Cuernavaca
  - Distrito Federal
  - Durango
  - Guadalajara
  - León
  - Mexico City
  - Monterrey
  - Oaxaca City
  - Veracruz
  - Zamora
- New Zealand (5):
  - Christchurch
  - Grafton
  - Hamilton
  - Palmerston North
  - Wellington
- Poland (5):
  - Gdansk
  - Lodz
  - Opole
  - Otwock
  - Wroclaw
- Puerto Rico (2):
  - Ponce
  - San Juan
- Romania (4):
  - Brasov
  - Bucharest
  - Cluj-Napoca
  - Iași
- Russia (12):
  - Barnaul
  - Kazan'
  - Moscow
  - Nizhny Novgorod
  - Obninsk
  - Omsk
  - Pyatigorsk
  - Rostov-on-Don
  - Saint Petersburg
  - Stavropol
  - Ufa
  - Yekaterinburg
- Singapore, Singapore
- South Korea (3):
  - Hwasun Gun
  - Seongnam-Si, Gyeonggi-Do
  - Seoul
- Spain (13):
  - A Coruña
  - Badajoz
  - Barakaldo Vizcaya
  - Barcelona
  - Córdoba
  - Hospitalet. Barcelona
  - Madrid
  - Palma de Mallorca
  - Salamanca
  - Santa Cruz de Tenerife
  - Seville
  - Toledo
  - Valencia
- Taiwan (3):
  - Kaohsiung City
  - Kaohsiung County
  - Taoyuan District
- Bangkok, Thailand

REFERENCES:
- [Derived] Sternberg CN, Castellano D, Daugaard G, Geczi L, Hotte SJ, Mainwaring PN, Saad F, Souza C, Tay MH, Garrido JM, Galli L, Londhe A, De Porre P, Goon B, Lee E, McGowan T, Naini V, Todd MB, Molina A, George DJ; Abiraterone Global EAP Investigators. Abiraterone acetate for patients with metastatic castration-resistant prostate cancer progressing after chemotherapy: final analysis of a multicentre, open-label, early-access protocol trial. Lancet Oncol. 2014 Oct;15(11):1263-8. doi: 10.1016/S1470-2045(14)70417-6. Epub 2014 Sep 18. PMID 25242048
- See also: An Open-Label Study of Abiraterone Acetate in Subjects with Metastatic Castration-Resistant Prostate Cancer Who Have Progressed After Taxane-Based Chemotherapy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=867&filename=CR017479_CSR.pdf